CLINICAL TRIAL: NCT00845130
Title: Quantitative in Vivo Biomarkers of Oxidative Stress in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: In-Young Choi, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, In-Young Choi, Ph.D., Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11119
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes; Oxidative Stress
Keywords: Diabetes; MR imaging; Vitamin C
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetic Type II Subjects (Experimental): Subjects received ascorbic acid (Vitamin C) infusion 1 g/kg (maximum 100gm
  Interventions: Biological: ascorbic acid (Vitamin C)
- Healthy Subjects (Experimental): Subjects received ascorbic acid (Vitamin C) infusion 1 g/kg (maximum 100gm
  Interventions: Biological: ascorbic acid (Vitamin C)

INTERVENTIONS:
Biological: ascorbic acid (Vitamin C) — ascorbic acid IV 1 g/kg
  Other Names: Vitamin C

SUMMARY:
Oxidative stress has been implicated in the development and complications of diabetes. Hyperglycemia and insulin resistance or insufficiency in diabetes can cause oxidative stress by excessive reactive oxygen species and can increase damage and alter antioxidant status in nerve cells. Antioxidant defense mechanisms protect against damage or restore oxidative damage. Glutathione, a powerful antioxidant plays a key role in the first line of antioxidant defense and seems to be a sensitive indicator of oxidative stress in various diseases such as diabetes. Glutathione functions in the regeneration of vitamin C which is another crucial antioxidant. Both hyperglycemia and insulin insufficiency inhibit uptake of vitamin C. The brain contains measurable amounts of glutathione that contribute to the antioxidant pool in the brain and guards against disease processes that are caused by oxidative stress. Since the brain is the most highly oxidative organ in the body and highly susceptible to oxidative stress, with increasing impact on diabetes, biomarkers of oxidative stress in the brain through the use of novel magnetic resonance imaging techniques for glutathione and vitamin C will be studied.

DETAILED DESCRIPTION:
The brain contains measurable amounts of glutathione that contribute to the antioxidant pool in the brain and guards against disease processes that are caused by oxidative stress. Since the brain is the most highly oxidative organ in the body and highly susceptible to oxidative stress, with increasing impact on diabetes, biomarkers of oxidative stress in the brain through the use of novel magnetic resonance imaging techniques for glutathione and vitamin C will be studied.

ELIGIBILITY:
Inclusion Criteria:

* 30-55 years of age
* Diabetic being treated with diet and any of the following: insulin, or other diabetic specific drug such as metformin, sulfonylurea or sitagliptin.
* Healthy subjects age and gender matched to diabetes patient

Exclusion Criteria:

* Use of any anti-inflammatory or antioxidant medications other than small daily doses of Aspirin (ASA:325 mg) and a daily multivitamin
* Co-existing chronic inflammatory conditions such as Crohn's disease, rheumatoid arthritis, chronic or acute infections
* Any concurrent neurological disease except for mild diabetic autonomic or peripheral neuropathy
* Postmeal C peptide > 0.3 mg/dl
* Normal healthy subjects who have any abnormal inflammatory marker, hyperlipidemia, or concurrent disease
* Diseases associated with abnormal glutathione metabolism
* Elevated serum creatinine levels, abnormal complete blood count (CBC), abnormal liver function tests or elevated serum homocysteine
* Morbid obesity
* History of hypoglycemic unawareness
* Pregnant women and women who are breastfeeding
* Patients with poor venous access
* Smokers
* Subject who consumes an excess of alcohol or abuses drugs
* History or or presence of bleeding disorder or use of anticoagulant drug
* History of oxalate renal calculi

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In-Young Choi, PhD, Principal Investigator — Un iversity of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
No, there is not a plan to share individual data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were consented to participate in the study. After baseline information was gathered from labs, it was determined that seven subjects did not meet the inclusion criteria. They were excluded from completing the study.
Groups:
- Diabetic Type II Subjects; Healthy Subjects: Subjects received ascorbic acid (Vitamin C) infusion 1 g/kg (maximum 100gm).
Period: Overall Study
Arm/Group | Diabetic Type II Subjects | Healthy Subjects
Started | 20 | 22
Completed | 16 | 19
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Health Subjects: Subjects received ascorbic acid (Vitamin C) infusion 1 g/kg (maximum 100gm).
- Total: Total of all reporting groups
Arm/Group | Diabetic Type II Subjects | Health Subjects | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (5) | 45 (7) | 47 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Vitamin C in Type 2 Diabetic Patients.
Description: Concentrations of vitamin C were measured in the brains of type 2 Diabetic patients and healthy controls.
Time Frame: Pre-Vitamin C infusion
Population: Determine cerebral concentrations of vitamin C. Data from one healthy subject were not usable due to subject's movement during MRI scan.
Measure: Mean (Standard Deviation); unit: umol/g tissue
Groups:
- Diabetic Type II Subjects: Vitamin C level in the living brain
- Healthy Subjects: Vitamin C levels in the living brain.
Arm/Group | Diabetic Type II Subjects | Healthy Subjects
Number analyzed (Participants) | 16 | 18
umol/g tissue | 1.1 (0.2) | 1.2 (0.1)

2. Primary Outcome: Quantify the Effect of Chronic Hyperglycemia on Cellular Uptake of Vitamin C Across the Blood-brain Barrier
Description: Concentrations of vitamin C after IV infusion of Vitamin C were measured in the brains of patients with type 2 diabetes and healthy controls to examine whether the concentrations are different between two groups.
Time Frame: 2 hour post infusion
Population: Data from one healthy subject were not usable due to subject's movement during MRI scan.
Measure: Mean (Standard Deviation); unit: µmol/g tissue
Arm/Group | Diabetic Type II Subjects | Healthy Subjects
Number analyzed (Participants) | 16 | 18
µmol/g tissue | 1.1 (0.2) | 1.4 (0.2)

ADVERSE EVENTS:
Arm/Group | Diabetic Type II Subjects | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No